CLINICAL TRIAL: NCT00729144
Title: Adaptive Behaviors Among Women With Bowel Incontinence: The ABBI Trial
Acronym: ABBI
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Office of Research on Women's Health (ORWH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Susan Meikle, MD, NICHD
Other Study IDs: 1J06-FI; U01HD041249 (NIH); U10HD041250 (NIH); U10HD041261 (NIH); U10HD041267 (NIH); U10HD054136 (NIH); U10HD054214 (NIH); U10HD054215 (NIH); U10HD054241 (NIH)
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-10

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; bowel incontinence; pelvic floor disorder
MeSH Terms: conditions — Fecal Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study focuses on the validation of the Adaptation Index instrument as a measurement of adaptive behaviors used to reduce symptoms of FI and to describe the use of adaptive behaviors among women with FI.

DETAILED DESCRIPTION:
It is common knowledge that women with pelvic floor dysfunction will develop, initiate and adopt behaviors which mitigate their symptoms or impairment. For some women, this involves wearing a pad and for others, knowledge of restroom locations. Little is known about the role of such behaviors in helping women adapt to urinary incontinence (UI), pelvic organ prolapse (POP), or fecal incontinence (FI). Additionally, there are no studies that address the persistence of these behaviors following treatment as measured by traditional outcomes. Results of a pilot study that assessed quality of life (QOL) in women with pelvic floor disorders (PFD) indicated that women relied heavily on behavioral adaptation in order to cope with PFD symptoms. Subsequently, a draft Adaptation Index was developed with input from investigators of the Pelvic Floor Disorders Network (PFDN). This measure was further refined by focus groups as part of the 1J06 protocol. The 1J06 study is investigating the properties of this tool in subjects with UI and POP. This study focuses on the validation of this instrument as a measurement of adaptive behaviors used to reduce symptoms of FI and to describe the use of adaptive behaviors among women with FI.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of FI with liquid, solid stool, or mucous incontinence, occurring at least monthly for 3 consecutive months. These women are planning to have treatment for FI.
* Women with prior treatment, including surgery for their FI, UI, and/or POP may be included if they now have a primary complaint of FI as defined above and are planning to have additional or new treatment for FI.

Exclusion Criteria:

* Diagnosis of interstitial cystitis, , bladder or colo-rectal malignancy or inflammatory bowel disease
* Refusal or inability to provide written consent
* Inability to complete telephone interviews conducted in English or Spanish
* Prior pelvic irradiation
* Incontinence only to flatus
* Prior removal of any portion of the colon or rectum
* Current or history of rectovaginal fistula(e)
* Rectal prolapse
* Neurologic disorders known to affect continence, including Multiple Sclerosis, Spinal Cord Injury, Debilitating Stroke, and Parkinson's Disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: women with a primary complaint of FI (with or without UI or POP) who are seeking treatment
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Adaptation Index and domains | baseline, 2 wk, 3 mo, 12 mo

SECONDARY OUTCOMES:
Fecal Incontinence Severity Index (FISI) | baseline, 2 wk, 3 mo, 12 mo
Medical Outcome Study Short-Form (SF-12) | baseline, 3 mo, 12 mo
Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ) | baseline, 3 mo, 12 mo
Modified Manchester Health Questionnaire | baseline, 3 mo, 12 mo
Patient Global Impression of Improvement (PGI-I) | 3 mo, 12 mo

CONTACTS AND LOCATIONS:
Overall Officials: Holly E Richter, PhD, MD, Study Chair — The University of Alabama at Birmingham; Alayne Markland, MD, Study Chair — The University of Alabama at Birmingham
Locations (8):
- United States (8):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego Medical Center, La Jolla, California
  - Kaiser Permanente, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Jelovsek JE, Chen Z, Markland AD, Brubaker L, Dyer KY, Meikle S, Rahn DD, Siddiqui NY, Tuteja A, Barber MD. Minimum important differences for scales assessing symptom severity and quality of life in patients with fecal incontinence. Female Pelvic Med Reconstr Surg. 2014 Nov-Dec;20(6):342-8. doi: 10.1097/SPV.0000000000000078. PMID 25185630
- [Derived] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495